CLINICAL TRIAL: NCT01310777
Title: Safety and IOP-Lowering Efficacy of Brinzolamide 10 mg/mL/Brimonidine 2 mg/mL Fixed Combination Eye Drops, Suspension Compared to Brinzolamide 10 mg/mL Eye Drops, Suspension and Brimonidine 2 mg/mL Eye Drops, Solution in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Brinzolamide/Brimonidine Twice a Day (BID) Fixed Combination (FC) vs Brinzolamide BID and Brimonidine BID in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-040; 2010-024512-34 (EudraCT Number)
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2013-12

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle glaucoma; Ocular Hypertension; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brinz/Brim (Experimental): Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension, 1 drop instilled in each eye 2 times a day for 6 months
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
- Brinz (Active Comparator): Brinzolamide 1% ophthalmic suspension, 1 drop instilled in each eye 2 times a day for 6 months
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension
- Brim (Active Comparator): Brimonidine tartrate 0.2% ophthalmic solution, 1 drop instilled in each eye 2 times a day for 6 months
  Interventions: Drug: Brimonidine tartrate 0.2% ophthalmic solution

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% ophthalmic suspension
  Arms: Brinz/Brim
Drug: Brinzolamide 1% ophthalmic suspension
  Other Names: AZOPT™
  Arms: Brinz
Drug: Brimonidine tartrate 0.2% ophthalmic solution
  Arms: Brim

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of Brinzolamide/Brimonidine in lowering intraocular pressure (IOP) relative to each of its individual active components in patients with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of 7 visits conducted during 2 sequential phases: the screening/eligibility phase, which included a screening visit and 2 eligibility visits, and a treatment phase, which included 4 on-therapy visits conducted at Week 2, Week 6, Month 3, and Month 6 (or early exit). Following washout of any IOP-lowering medication, subjects who met all inclusion/exclusion criteria at both eligibility visits and who had IOP measurements within the specified range during this period were randomized to 1 of 3 study drug groups: Brinz/Brim, Brinz, or Brim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open angle glaucoma or ocular hypertension, and, in the opinion of the Investigator, are insufficiently controlled on monotherapy or are currently on multiple IOP-lowering medications.
* Meet qualifying IOP entry criteria.
* Able to understand and sign an informed consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, test positive for pregnancy at Screening Visit, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Severe central visual field loss.
* Best corrected visual acuity (BCVA) score worse than 55 ETDRS letters (20/80 Snellen equivalent).
* Chronic, recurrent or severe inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or ocular inflammation within the preceding 3 months.
* Clinically significant or progressive retinal disease.
* Other ocular pathology.
* Intraocular surgery within the 6 months prior to entry.
* Ocular laser surgery within the 3 months prior to entry.
* Any abnormality preventing reliable applanation tonometry.
* Any other conditions, including severe illness, which would make the subject, in the opinion of the Investigator, unsuitable for the study.
* Recent use of high-dose (>1 gram daily) salicylate therapy.
* Recent, current, or anticipated treatment with any medication that augments adrenergic responses, or precludes use of an alpha-adrenergic agonist.
* Concurrent use of glucocorticoid medications administered by any route.
* Other protocol-specified exclusion crtieria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 771 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Teague, Sr. Clinical Manager, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 63 investigational centers in the Asia-Pacific region, the European Union, Latin America and Caribbean nations, and the United States.
Pre-assignment Details: Of the 771 enrolled, 211 subjects did not meet inclusion/exclusion criteria and were exited from the study as screen failures prior to randomization. This reporting group includes all randomized subjects (560).
Period: Overall Study
Arm/Group | Brinz/Brim | Brinz | Brim
Started | 193 | 192 | 175
Completed | 160 | 178 | 145
Not Completed | 33 | 14 | 30
Not completed — Adverse Event | 23 | 1 | 15
Not completed — Lost to Follow-up | 0 | 4 | 1
Not completed — Patient's Decision Unrelated to AE | 1 | 1 | 2
Not completed — Inadequate Control of IOP | 5 | 7 | 10
Not completed — Other | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: This reporting group includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinz | Brim | Total
Number analyzed (Participants) | 193 | 192 | 175 | 560
Age, Customized [Number; unit: participants]
  <65 years | 91 | 87 | 79 | 257
  ≥65 years | 102 | 105 | 96 | 303
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 102 | 102 | 310
  Male | 87 | 90 | 73 | 250

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP Change From Baseline at Month 3
Description: Mean Diurnal IOP Change from Baseline at Month 3 (ie, the subject IOP change from baseline averaged over the 9 AM, + 2 h, and + 7 h time points at Month 3) was measured by Goldmann applanation tonometry. The study drug was instilled approximately 15 minutes after conducting the 9AM IOP measurement. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Baseline (Day 1), Month 3
Population: The intent-to-treat (ITT) analysis set included all subjects who received study drug and completed at least 1 scheduled on-therapy study visit.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Brinz/Brim | Brinz | Brim
Number analyzed (Participants) | 176 | 182 | 161
millimeters of mercury (mmHg) | -7.9 (0.22) | -6.5 (0.23) | -6.4 (0.24)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (1 year, 8 months). An AE was defined as any untoward medical occurrence in a subject who was administered a study medication, regardless of causal relationship with the medication.
Description: This reporting group includes all subjects exposed to study drug. Reports of AEs were obtained through solicited and spontaneous comments from the study subjects, and through observations by the study Investigator as outlined in the study protocol.
Arm/Group | Brinz/Brim | Brinz | Brim
Serious Adverse Events (participants affected / at risk) | 5/193 | 2/192 | 3/175
Other Adverse Events (participants affected / at risk) | 44/193 | 12/192 | 18/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=193) | Brinz (N=192) | Brim (N=175)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=193) | Brinz (N=192) | Brim (N=175)
Ocular hyperaemia (Eye disorders) | 11 | 3 | 9
Conjunctivitis (Eye disorders) | 11 | 2 | 2
Vision Blurred (Eye disorders) | 11 | 1 | 3
Eye Pain (Eye disorders) | 11 | 3 | 0
Dry Mouth (Gastrointestinal disorders) | 7 | 2 | 9
Dysgeusia (Nervous system disorders) | 11 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.